CLINICAL TRIAL: NCT02900560
Title: Phase II Randomized Study of Pembrolizumab With or Without Epigenetic Modulation With CC-486 in Patients With Platinum-resistant Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Study of Pembrolizumab With or Without CC-486 in Patients With Platinum-resistant Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research in Oncology (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIO026
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — cc-486; Azacitidine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Active Comparator): CC-486 100 mg once a day, 21 days on, 7 days off combined with Pembrolizumab 200 mg IV every 21 days
  Interventions: Drug: CC-486; Biological: Pembrolizumab
- Cohort 2 (Active Comparator): CC-486 100 mg twice a day, 21 days on, 7 days off combined with Pembrolizumab 200 mg IV every 21 days
  Interventions: Drug: CC-486; Biological: Pembrolizumab
- Cohort 3 (Active Comparator): CC-486 300 mg once a day, 14 days on and 14 days off combined with Pembrolizumab 200 mg IV every 21 days
  Interventions: Drug: CC-486; Biological: Pembrolizumab
- Cohort 4 (Active Comparator): CC-486 300 mg once a day, 21 days on, 7 days off combined with Pembrolizumab 200 mg IV every 21 days
  Interventions: Drug: CC-486; Biological: Pembrolizumab

INTERVENTIONS:
Drug: CC-486 — CC-486 Intervention will depend on cohort enrolled in. 100 mg tablet
  Other Names: oral azacitidine
Biological: Pembrolizumab — Pembrolizumab 200 mg IV every 21 days
  Other Names: Keytruda

SUMMARY:
The purpose of the study is to determine the optimal dose of CC-486 (oral azacitidine) in combination with pembrolizumab for the treatment of platinum-resistant/refractory Epithelial Ovarian Cancer (EOC).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, four-cohort study, in which intravenous pembrolizumab will be combined with 4 different schedules of administration of CC-486 (oral azacitidine), for the treatment of platinum-resistant/refractory (EOC). This is also a futility trial for the strategy to combine pembrolizumab and CC-486 in EOC. Eligible subjects will be treated in one of four cohorts of combined oral CC-486 and intravenous pembrolizumab (200 mg intravenous (IV) every 3 weeks in all cohorts) to evaluate the safety of each combination schedule and to have preliminary data on their efficacy. The primary objective is to establish the optimal dosing schedule for comparison with pembrolizumab alone.

Subjects will be assigned to a treatment cohort in the order they are enrolled in the study. In all subjects, tumor tissue will be obtained via image-guided core biopsy at study entry and 6 weeks after commencing treatment with CC-486. A cohort will remain open to accrual until five subjects treated on that cohort have completed two CC-486 cycles and have had the first post-baseline tumor burden assessment and both tumor biopsies performed and adequate paired tissue obtained. At least 5 evaluable subjects per cohort will be accrued over an estimated period of approximately 24 months.

Subjects will be treated in the assigned cohort until progressive disease based on Immune-Related Response Evaluation Criteria In Solid Tumors (irRECIST), unacceptable toxicity, consent withdrawal or the Investigator concludes that it is in the subject´s best interest to discontinue. Once 5 subjects in each cohort are considered evaluable for response, toxicity and treatment responses will be analyzed for each of the four cohorts and an optimal schedule will be selected.

This study includes mandatory tumor core biopsies for biomarkers research and mandatory whole blood sampling for deoxyribonucleic acid (DNA) methylation analyses.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent document obtained prior to initiation of any study-specific procedure and treatment (by the subject or a legally acceptable representative as per the local regulations).
* Women ≥ 18 years old
* Histologically confirmed Epitheilial Ovarian Cancer (EOC), Fallopian Tube Cancer (FTC) or Primary Peritoneal Cancer (PPC).
* Received debulking surgery and preoperative and/or postoperative platinum-based frontline chemotherapy (intravenous and/or intraperitoneal) for the treatment of EOC/FTC/PPC.
* Documented platinum-resistant or platinum-refractory disease. Platinum-resistant disease is defined as progression within < 6 months from completion of a minimum of 4 platinum frontline therapy cycles in the pre or postoperative setting (the date should be calculated from the last administered dose of platinum agent). Platinum-refractory is defined as disease that has recurred/progressed while receiving platinum-based frontline therapy.
* Measurable disease according to Immune-Related Response Evaluation Criteria In Solid Tumors (irRECIST)
* Indication of systemic treatment for the relapsed EOC, FTC or PPC.
* Subjects must have a tumor lesion that is amenable to an image-guided core biopsy and willingness to undergo two biopsies (baseline and 6 weeks after first dose of study treatment).
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0 or 1.
* Expected survival of more than 6 months.
* Adequate organ function within 7 days prior to enrollment, as defined by the following criteria:

  * Absolute neutrophils count (ANC) ≥ 1.5 x 10E9/L, platelets ≥ 100 x 10E9/L, hemoglobin > 9 g/dL (without transfusion or erythropoiesis stimulating agents' dependency).
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN).
  * Total serum bilirubin ≤ 1.5 x ULN regardless of liver involvement secondary to tumor. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
  * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) < 2.0 x ULN or ≤ 5 X ULN for subjects with liver metastases.
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Partial Thromboplastin Time (PTT) or Activated Partial Thromboplastin Time (aPTT) ≤ 40 seconds unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* For women of childbearing potential, negative serum pregnancy test within 7 days of enrollment
* Women of childbearing potential must agree to use acceptable methods of birth control starting with the screening visit and up to 120 days after the last dose of study treatment. Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Non-epithelial ovarian cancers, including malignant mixed Müllerian tumors.
* Ovarian tumors with low malignant potential (i.e. borderline tumors).
* Relapse/progression based solely on elevation of CA-125, in absence of measurable disease, according to irRECIST criteria.
* More than 2 prior treatment regimens for the platinum-resistant/refractory relapsed EOC, FTC, or PTC, defined as investigational, chemotherapy, hormonal, biologic, or targeted therapy.
* Any concurrent or previous malignancy within 5 years prior to enrollment except for adequately and radically treated basal or squamous skin cancer, or carcinoma in situ of the cervix, or other non-invasive/in-situ neoplasm. A subject with previous history of invasive malignancy (other than adequately and radically treated basal or squamous skin cancer or carcinomas in situ) is eligible provided that she has been disease free for more than 5 years.
* Brain metastases (even if treated and/or stable), spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.
* Prior systemic anticancer therapy within 4 weeks prior to enrollment or who has not recovered (i.e. ≤ Grade 1 or baseline grade) from adverse events due to a previously administered agent
* Prior treatment with a monoclonal antibody within 4 weeks prior to enrollment or who has not recovered (i.e. ≤ Grade 1 or baseline grade) from adverse events due to agents administered more than 4 weeks earlier.
* Diagnosis of immunosuppression or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment . The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor.
* Active autoimmune disease or history of autoimmune disease or syndrome that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects with vitiligo or resolved childhood asthma/atopy will not be excluded.
* Received live vaccines within 30 days prior to enrollment
* Current or prior history of myelodysplastic syndrome, leukemia or clinically significant (as per Investigator judgment) bone marrow failure.
* Uncontrolled systemic fungal, bacterial or viral infection at time of enrollment (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment).
* Known history of active TB (Bacillus Tuberculosis).
* Known HIV infection or known history of Hepatitis B or known positivity for active Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative] is detected).
* Known history of non-infectious pneumonitis that required steroids or has current pneumonitis (infectious or non-infectious).
* Significant active cardiac disease within 6 months prior to enrollment, including but not limited to New York Heart Association class 4 cardiac heart failure, unstable angina, myocardial infarction
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator. Is or has an immediate family member (e.g. spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
* Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Prior treatment with any anti-Programmed Death (PD)-1, or PD-L1 or PD-L2 agent; or with azacitidine (any formulation) or any other hypomethylating agent; or with anti-cytoplasmic (CD) 137, or anti-cytotoxic T-Lymphocyte Associated Protein (CTLA)-4 antibody (including ipilimumab) or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Known or suspected hypersensitivity to azacitidine, pembrolizumab or the excipients of any of the study drugs (including mannitol). Known or suspected hypersensitivity to monoclonal antibodies.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks prior to enrollment .
* Pregnant or lactating women or is expecting to conceive children or breastfeed within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Fresco, MD, Study Director — Translational Research in Oncology
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 10 | 7 | 8
Completed | 7 | 10 | 7 | 8
Not Completed | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 9 | 10 | 7 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (8.89) | 59.9 (13.15) | 63.7 (12.47) | 68.0 (6.39) | 62.2 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 7 | 8 | 34
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 10 | 6 | 7 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Primary Tumor Location [Count of Participants; unit: Participants]
  Epithelial Ovarian Cancer | 7 | 9 | 6 | 4 | 26
  Fallopian Tube Carcinoma | 1 | 0 | 1 | 4 | 6
  Primary Peritoneal Carcinoma | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3, 4, or 5 Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Description: Safety evaluation: number of subjects with grade 3, 4, or 5 adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. This is an assessment of the frequency, severity and relationship to trial treatment of all adverse events that occurred while on trial. CTCAE is a standard classification and severity grading scale (from 1- mild to 5 - death) for adverse events in clinical trials and oncology settings.
Time Frame: The average time period for patient participation was 30 weeks.
Population: Analysis is completed using the Safety Population as opposed to the "Intent-to-Treat" Population (all patients who were enrolled in the study, regardless of whether they actually received study medication). The Safety Population consists of all patients who receive any study treatment, and will be used for the analysis of safety data of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 10 | 7 | 8
Participants
  Patients with any Grade 3 or 4 Adverse Event | 5 | 8 | 5 | 7
  Patients with Grade 5 Adverse Event | 1 | 0 | 0 | 0
  Patients without Grade 3, 4, or 5 Adverse Event | 1 | 2 | 2 | 1

2. Primary Outcome: Number of Subjects With Immune-related Partial Response (irPR), Immune-related Complete Response (irCR), Immune-related Stable Disease (irSD), Immune-related Progressive Disease (irPD), and Immune-related Not Evaluable (irNE) as Assessed by irRECIST.
Description: Efficacy evaluation: based on the Immune-related Objective Response Rate (irORR)/ Immune-related Disease Control Rate (irDCR) per Immune-Related Response Evaluation Criteria In Solid Tumor (irRECIST) criteria using the intent-to-treat (ITT) population (all patients who were enrolled in the study, regardless of whether they actually received study medication). The best overall response outcome (irCR/irPR/irSD/irPD/irNE) will be summarized and tabulated for ITT by cohort.
Time Frame: The average time period for patient participation was 30 weeks.
Population: Analysis was performed on the intent-to-treat (ITT) population (i.e., patients who were enrolled in the study, regardless of whether they actually received study medication), which is different from the safety population (i.e., patients who receive any study treatment) used for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 9 | 10 | 7 | 8
Participants
  irPR | 0 | 0 | 1 | 0
  irCR | 0 | 0 | 0 | 0
  irSD | 3 | 6 | 3 | 4
  irPD | 5 | 2 | 1 | 4
  irNE | 0 | 1 | 0 | 0
  Missing | 1 | 1 | 2 | 0

3. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events Related to CC-486 as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Description: Safety evaluation: number of subjects with treatment emergent adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. This is an assessment of the frequency and relationship to trial treatment of all adverse events that occurred while on trial. CTCAE is a standard classification and severity grading scale (from 1- mild to 5 - death) for adverse events in clinical trials and oncology settings.
Time Frame: The average time period for patient participation was 30 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 10 | 7 | 8
Participants | 7 | 10 | 7 | 8

4. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events Related to Pembrolizumab as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Description: as for outcome 3
Time Frame: The average time period for patient participation was 30 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 10 | 7 | 8
Participants | 6 | 5 | 6 | 3

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected the from the time when the first patient consented (signed informed consent form) to the end of study for the last patient. The average timeframe for patient participation was 30 weeks for which data was collected/assessed.
Description: The SAFETY population was used to assess clinical safety and tolerability and consisted of all subjects who were enrolled (Part A) and received at least one dose of study medication (this is different from the intent-to-treat population, which included all patients enrolled in the study, irrespective of treatment). All adverse experiences observed by the Investigator or reported by the patient were collected at each visit and any contact during the study and follow-up period.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 6/7 | 4/10 | 1/7 | 3/8
Serious Adverse Events (participants affected / at risk) | 3/7 | 6/10 | 3/7 | 1/8
Other Adverse Events (participants affected / at risk) | 7/7 | 10/10 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=10) | Cohort 3 (N=7) | Cohort 4 (N=8)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=10) | Cohort 3 (N=7) | Cohort 4 (N=8)
Vomiting (Gastrointestinal disorders) | 5 | 6 | 7 | 8
Nausea (Gastrointestinal disorders) | 5 | 7 | 5 | 7
Constipation (Gastrointestinal disorders) | 7 | 4 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 4 | 7
Abdominal Pain (Gastrointestinal disorders) | 2 | 3 | 1 | 1
Ascites (Gastrointestinal disorders) | 3 | 1 | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 6 | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 6 | 7
Pyrexia (General disorders) | 4 | 1 | 1 | 0
Odema Peripheral (General disorders) | 1 | 1 | 1 | 1
Chills (General disorders) | 1 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Early satiety (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 2 | 5
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 2 | 2 | 2
Weight decreased (Investigations) | 2 | 1 | 1 | 3
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 3
Platelet count decreased (Investigations) | 1 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 1 | 6 | 4
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Trial closed prematurely with 34 participant enrolled in Part A of the study. All of the treatment cohorts met at least one of the safety rejection criteria. Enrollment took 31 months, significantly longer than anticipated (24 months).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication, abstract or presentation of the study will be made without the approval of the Study Steering Committee (SSC).

DOCUMENTS (2):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT02900560/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02900560/SAP_001.pdf